CLINICAL TRIAL: NCT04991480
Title: A Phase I/IIa, Open-label, Multi-centre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of the DNA Polymerase Theta Inhibitor ART4215 Administered Orally as Monotherapy and in Combination to Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of ART4215 for the Treatment of Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Artios Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ART4215C001
Record Dates: First submitted 2021-07-19; First posted 2021-08-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Advanced Cancer; Metastatic Cancer; Breast Cancer
Keywords: Sensitivity to pol theta inhibition; Germline Breast Cancer gene mutation; gBRCA-m; BRCA1; BRCA2; Human epidermal growth factor receptor 2 negative; HER2 negative
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms | interventions — talazoparib; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A1 (Experimental): Part A1 will evaluate ART4215 monotherapy administered in 21 day cycles. Up to 90 participants will participate in this dose escalation arm.
  Interventions: Drug: ART4215
- Part A2 (Experimental): Part A2 will evaluate ART4215 given in combination with talazoparib in 21 day cycles. Up to 50 participants will participate in this dose escalation arm.
  Interventions: Drug: ART4215; Drug: Talazoparib
- Part B1 (Experimental): In Part B1 dose expansion, up to 30 participants with solid cancers that have been treated with a PARP inhibitor for an approved indication will receive ART4215.
  Interventions: Drug: ART4215
- Part B2 (Experimental): In Part B2 dose expansion, up to 20 participants with solid cancers with characteristics indicative of sensitivity to pol theta inhibition will receive ART4215.
  Interventions: Drug: ART4215
- Part B3 (Experimental): In Part B3, approximately 120 participants with HER2 negative BRCA breast cancers will be randomized 1:1 to either ART4215 in combination with talazoparib or talazoparib alone.
  Interventions: Drug: ART4215; Drug: Talazoparib
- Part A3 (Experimental): Part A3 will evaluate ART4215 given in combination with niraparib in 21-day cycles. Up to 30 participants will participate in this dose escalation arm.
  Interventions: Drug: ART4215; Drug: Niraparib

INTERVENTIONS:
Drug: ART4215 — Participants will receive ART4215 by mouth daily in 21-day cycles.
Drug: Talazoparib — Talazoparib will be administered at a dose of 1 mg or 0.75 mg by mouth daily in 21-day cycles.
  Other Names: Talzenna
  Arms: Part A2; Part B3
Drug: Niraparib — Niraparib will be administered at a dose of 200 mg or 300 mg by mouth daily in 21-day cycles.
  Other Names: Zejula
  Arms: Part A3

SUMMARY:
This clinical trial is evaluating a drug called ART4215 in participants with advanced or metastatic solid tumors. The main goals of this study are to:

* Find the recommended dose of ART4215 that can be given safely to participants alone and in combination with talazoparib
* Learn more about the side effects of ART4215 alone and in combination with talazoparib
* Learn more about the effectiveness of ART4215 alone and in combination with talazoparib
* Learn more about the effectiveness of ART4215 alone and in combination with niraparib

DETAILED DESCRIPTION:
This is an open-label Phase I/IIa study designed to evaluate ART4215, a new first-in-class investigational medicinal product that is a potent and selective inhibitor of deoxyribonucleic acid (DNA) polymerase (pol) theta. ART4215 is being developed as an oral anti-cancer agent for monotherapy treatment of patients with cancers that harbor defects in DNA repair and in combination with anticancer medicines that cause DNA damage.

This study was intended to be a Phase I/IIa trial, however the trial did not proceed to the Phase IIa portion of the study.

ELIGIBILITY:
General Inclusion Criteria:

* Signed informed consent
* Discontinued all previous treatments for cancer for at least 21 days or 5 half-lives, whichever is shorter (except in Germany where local regulation requires the longer of 21 days or 5 half-lives washout), and recovered from the acute effects of therapy. Palliative radiotherapy must have completed 1 week prior to start of study treatment.
* At least 1 radiologically evaluable lesion (measurable and/or non-measurable) that can be assessed at baseline and is suitable for repeated radiological evaluation by RECIST v1.1 or Prostate Cancer Working Group-3 (PCWG-3) for patients with prostate cancer
* Acceptable hematologic, renal, hepatic, and coagulation functions independent of transfusions and granulocyte colony-stimulating factor
* Willingness to abide by protocol defined contraceptive requirements for the duration of the study.
* Estimated life expectancy of ≥12 weeks

Additional inclusion criteria for participants in dose escalation (Part A1):

* Advanced or metastatic cancer, which is refractory to standard therapies, or for which no standard therapies exist, or for which the investigator feels no other active therapy is required for the duration of the study
* Non-irradiated tumor tissue sample (archival or newly obtained core biopsy of a tumor lesion) available for submission for analysis

Additional inclusion criteria for participants in dose escalation (Part A2):

* Advanced or metastatic cancer for which a PARP inhibitor is an appropriate treatment option. Participants may have received prior treatment with PARP inhibitor
* Optional baseline biopsy for BRCA1/2 mutations and prior PARP inhibitor
* Non-irradiated tumor tissue sample (archival or newly obtained core biopsy of a tumor lesion) available for submission for analysis

Additional inclusion criteria for participants in dose escalation (Part A3):

* Advanced or metastatic cancer for which a PARP inhibitor is an appropriate treatment option. Prior treatment with PARP inhibitor
* Non-irradiated tumor tissue sample (archival or newly obtained core biopsy of a tumor lesion) available for submission for analysis

Additional inclusion criteria for participants in dose expansion (Part B1):

* Advanced or metastatic solid tumors that have undergone disease progression during treatment with a PARP inhibitor for an approved indication
* At least 1 measurable lesion assessable using standard techniques by RECIST v1.1 or PCWG-3 guidelines
* Non-irradiated tumor tissue sample (archival or newly obtained core biopsy of a tumor lesion) available for submission for analysis

Additional inclusion criteria for participants in dose expansion (Part B2):

* Advanced or metastatic cancer that is refractory to standard therapies, or for which no standard therapies exist, or for which the investigator feels no other active therapy is required for the duration of the study with characteristics indicative of sensitivity to pol theta inhibition
* No prior treatment with a PARP inhibitor and must not have a disease for which there is an approved PARP inhibitor
* At least 1 measurable lesion assessable using standard techniques by RECIST v1.1 or PCWG-3 guidelines
* Non-irradiated tumor tissue sample (archival or newly obtained core biopsy of a tumor lesion) available for submission for analysis

Additional inclusion criteria for participants in dose expansion (Part B3):

* HER2-negative locally advanced or metastatic breast cancer
* Deleterious or suspected deleterious germline or somatic BRCA1 or BRCA2 mutation
* No more than 3 prior chemotherapy-inclusive regimens (including antibody conjugates)
* Prior treatment with a taxane or anthracycline unless contraindicated
* No or </= 1 month of prior treatment with a PARP inhibitor
* At least 1 measurable lesion assessable using standard techniques by RECIST v1.1
* Non-irradiated tumor tissue sample (archival or newly obtained core biopsy of a tumor lesion) available for submission for analysis

General Exclusion Criteria:

* Women who are pregnant, breast feeding, or who plan to become pregnant while in the study or within the protocol defined timeframe after the last administration of study specified treatment.
* Men who plan to father a child while in the study or within the protocol defined timeframe after the last administration of study specified treatment.
* Serious concomitant systemic disorder that would compromise the participants ability to adhere to the protocol including: opportunistic HIV/AIDs-related infection(s) within the past 12 months, hepatitis B virus, or hepatitis C virus; documented active or chronic tuberculosis infection; malignancy prior to the one currently being treated [including myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)] that is not in remission
* Have MDS/AML or features suggestive of MDS/AML
* Ongoing interstitial lung disease or pneumonitis (whether symptomatic or asymptomatic)
* Moderate or severe cardiovascular disease
* Symptomatic or uncontrolled brain metastases, spinal cord compression, or leptomeningeal disease requiring concurrent treatment; stable brain metastases are eligible
* Received a live vaccine within 30 days before the first dose of study treatment
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate
* Recent major surgery within 4 weeks prior to entry into the study or minor surgery within 1 week of entry into the study
* Significant bleeding disorder or vasculitis or had a Grade ≥3 bleeding episode within 12 weeks prior to enrollment
* Currently enrolled in a clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study

Additional exclusion criteria for participants in dose expansion (Part B3):

* First-line locally advanced and/or metastatic breast cancer with no prior adjuvant chemotherapy
* Inflammatory breast cancer
* Known hypersensitivity to any of the components of talazoparib
* Prior treatment with a PARP inhibitor that was discontinued due to a treatment related toxicity.

Additional exclusion criteria for participants in dose escalation (Part A3):

• Hypersensitivity to any of the components of niraparib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2025-12-24 (Actual)

PRIMARY OUTCOMES:
Part A: Number of participants with dose limiting toxicities (DLTs) from ART4215 monotherapy, in combination with talazoparib or in combination with niraparib | 21 days (Cycle 1)
  DLTs are defined as adverse events (graded according to NCI CTCAE v5.0) during Cycle 1 that are related to ART4215 monotherapy, in combination with talazoparib or in combination with niraparib
Part B1 and B2: Number of participants with adverse events following administration of ART4215 | From the first dose until up to 30 days after the last dose of ART4215. Each cycle is 21 days.
  Number of adverse events as characterized by type, frequency, seriousness (graded according to NCI CTCAE v5.0) and relationship to ART4215
Part B3: Progression free survival (PFS) as a measure of efficacy for ART4215 in combination with talazoparib or talazoparib alone | Every 6 weeks (±7 days) from date of randomization for 18 weeks, then every 9 weeks (±7 days) up to approximately 24 months. Each cycle is 21 days.
  PFS is defined as the time from the start of randomization until the earliest objective disease progression defined by RECIST v1.1 or death by any cause in the absence of progression.

SECONDARY OUTCOMES:
Part B3: Number of participants with adverse events following administration of ART4215 in combination with talazoparib | From the first dose until up to 30 days after the last dose of ART4215. Each cycle is 21 days.
  Number of adverse events as characterized by type, frequency, seriousness (graded according to NCI CTCAE v5.0) and relationship to ART4215 in combination with talazoparib
Best overall response (BOR) as a measure of efficacy for ART4215 as monotherapy, in combination with talazoparib or in combination with niraparib | Every 6 weeks (±7 days) from the first dose for 18 weeks, then every 9 weeks (±7 days) up to approximately 24 months. Each cycle is 21 days.
  BOR will be calculated as the best response from date study treatment started until progression or censoring date in the absence of progression. BOR will be based on RECIST v1.1 and Prostate Cancer Working Group-3 (PCWG-3) (for prostate cancer).
Objective response rate (ORR) as a measure of efficacy for ART4215 as monotherapy, in combination with talazoparib or in combination with niraparib | Every 6 weeks (±7 days) from the first dose for 18 weeks, then every 9 weeks (±7 days) up to approximately 24 months. Each cycle is 21 days.
  ORR is defined as the proportion of patients who have a best response of either complete response (CR) or partial response (PR) based on RECIST v1.1 or PCWG-3. Response must be confirmed (at least two responses of CR or PR a minimum of 4 weeks apart and prior to progression/subsequent therapy) for Parts A, B1 and B2.
Disease control rate (DCR) as a measure of efficacy for ART4215 as monotherapy, in combination with talazoparib or in combination with niraparib | Every 6 weeks (±7 days) from the first dose for 18 weeks, then every 9 weeks (±7 days) up to approximately 24 months. Each cycle is 21 days.
  DCR is defined as the proportion of patients with CR, PR, or SD based on RECIST v1.1 or PCWG-3.
Duration of response (DOR) as a measure of efficacy for ART4215 as monotherapy, in combination with talazoparib or in combination with niraparib | Every 6 weeks (±7 days) from the first dose for 18 weeks, then every 9 weeks (±7 days) up to approximately 24 months. Each cycle is 21 days.
  DOR will be defined for patients with a BOR of CR/PR as the time from the date of first documented response until date of documented progression (by RECIST v1.1 or PCWG-3) or death in the absence of disease progression. BOR should be confirmed in Parts A, B1, and B2.
Change in tumor size as a measure of efficacy for ART4215 as monotherapy, in combination with talazoparib or in combination with niraparib | Every 6 weeks (±7 days) from the first dose for 18 weeks, then every 9 weeks (±7 days) up to approximately 24 months. Each cycle is 21 days.
  Change in tumor size will be assessed for all patients with target lesion measurements at baseline.
Parts A, B1, and B2: Progression free survival (PFS) as a measure of efficacy for ART4215 as monotherapy, in combination with talazoparib or in combination with niraparib | Every 6 weeks (±7 days) from the first dose for 18 weeks, then every 9 weeks (±7 days) up to approximately 24 months. Each cycle is 21 days.
  PFS is defined as the time from the start of study treatment until the earliest objective disease progression defined by RECIST v1.1 or PCWG-3 or death by any cause in the absence of progression.
Overall survival (OS) as a measure of efficacy for ART4215 as monotherapy, in combination with talazoparib or in combination with niraparib | Assessed every 12 weeks after treatment discontinuation for up to 24 months.
  OS is defined as the time from the start of study treatment until death due to any cause.
Pharmacokinetic Analysis (single dose): maximum plasma concentration (Cmax) of ART4215 when given alone, in combination with talazoparib or in combination with niraparib | PK will be measured at each cycle from Cycle 0 to Cycle 3, and then every third cycle beginning at Cycle 5 for up to approximately 24 months. Each cycle is 21 days.
Pharmacokinetic Analysis (single dose): time to maximum plasma concentration (tmax) of ART4215 when given alone, in combination with talazoparib or in combination with niraparib | PK will be measured at each cycle from Cycle 0 to Cycle 3, and then every third cycle beginning at Cycle 5 for up to approximately 24 months. Each cycle is 21 days.
Pharmacokinetic Analysis (single dose): area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC(0-inf)) of ART4215 when given alone, in combination with talazoparib or in combination with niraparib | PK will be measured at each cycle from Cycle 0 to Cycle 3, and then every third cycle beginning at Cycle 5 for up to approximately 24 months. Each cycle is 21 days.
Pharmacokinetic Analysis (multiple dose): maximum plasma concentration (Cmax) of ART4215 when given alone, in combination with talazoparib or in combination with niraparib | PK will be measured at each cycle from Cycle 0 to Cycle 3, and then every third cycle beginning at Cycle 5 for up to approximately 24 months. Each cycle is 21 days.
Pharmacokinetic Analysis (multiple dose): time to maximum plasma concentration (tmax) of ART4215 when given alone, in combination with talazoparib or in combination with niraparib | PK will be measured at each cycle from Cycle 0 to Cycle 3, and then every third cycle beginning at Cycle 5 for up to approximately 24 months. Each cycle is 21 days.
Pharmacokinetic Analysis (multiple dose): area under the concentration-time curve over the dosing interval (AUC tau) of ART4215 when given alone, in combination with talazoparib or in combination with niraparib | PK will be measured at each cycle from Cycle 0 to Cycle 3, and then every third cycle beginning at Cycle 5 for up to approximately 24 months. Each cycle is 21 days.
Pharmacokinetic Analysis (single dose): maximum plasma concentration (Cmax) of ART4215 when given with or without food | 8 days (Cycle 0)
Part A2: Pharmacokinetic Analysis (multiple dose): maximum steady state plasma concentration (Cmax ss) of talazoparib when given in combination with ART4215 | 1 day (Cycle 2 Day 1; Cycle 2 is 21 days)
Pharmacokinetic Analysis (single dose): time to maximum plasma concentration (tmax) of ART4215 when given with or without food | 8 days (Cycle 0)
Pharmacokinetic Analysis (single dose): area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC(0-inf)) of ART4215 when given with or without food | 8 days (Cycle 0)
Assessment of lesions in (or indicative of lesions in) DNA repair pathways by immunohistochemistry for loss of shieldin complex and/or TP53BP1 or other relevant pathways | Within 28 days prior to the first dose of ART4215.
Pharmacokinetic Analysis (Part A1): renal clearance of ART4215 monotherapy will be calculated as the cumulative amount of ART4215 excreted unchanged in the urine (Ae) divided by the appropriate AUC. | PK will be measured on Cycle 0 Day -4 and Cycle 1 Day 8. Cycle 0 is 4 days. Cycle 1 is 21 days.
Pharmacokinetic Analysis (Parts A2/B3) : renal clearance of ART4215 in combination with talazoparib will be calculated as the cumulative amount of ART4215 excreted unchanged in the urine (Ae) divided by the appropriate AUC. | PK will be measured on Cycle 1 Day 1 and Cycle 1 Day 8. Cycle 1 is 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Hamilton, MD, Study Chair — Tennessee Oncology; Timothy Yap, MBBS, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (8):
- United States (7):
  - Yale School of Medicine, New Haven, Connecticut
  - Florida Cancer Specialists, Orlando, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oklahoma University, Oklahoma City, Oklahoma
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Sarah Cannon Research Institute, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No